CLINICAL TRIAL: NCT02452437
Title: Clinical Trial Simulation Using ODE/PDE Hemodialysis Model for Quantifying Oxycodone's Removal in End-Stage Kidney Disease
Brief Title: Opioids in Chronic Kidney Disease Patients Undergoing Hemodialysis
Acronym: OCKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Emerio & Lourdes Linares Research and Education Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ELLHDM-001
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Kidney Disease
Keywords: oxycodone; hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Experimental): Oxycodone will be administered and subjects will undergo hemodialysis
  Interventions: Drug: Oxycodone
- hemodialysis (Experimental): Oxycodone will be administered and subjects will undergo hemodialysis
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Controlled release oxycodone 40 mg twice daily
  Other Names: OxyContin

SUMMARY:
To measure oxycodone's intradialytic mass transfer rate coefficient and oxycodone's removal rate using an ODE/PDE hemodialysis model. To implement a rational clinical strategy for estimating a patient's post-hemodialysis oxycodone restoration dose using results from an ODE/PDE model of hemodialysis.

DETAILED DESCRIPTION:
Clinical Trial Simulation Design and Investigational Plan: Our study sample will consist of a group of 10 randomly selected virtual Caucasian hemodialysis patients with Stage 5 chronic kidney disease (CKD) and a group of 10 randomly selected Caucasian age and weight matched healthy controls. Patients, 5 women and 5 men in each group, will be synthesized using clinical trial simulation techniques from the case report data reported by Lee, Leng, and Cooper and the experiments by Kirvela and coworkers. Our goal is to learn about the populations from which the study samples are drawn. To meet this goal, the investigators will perform Monte Carlo simulation.

Both virtual control subjects and experimental hemodialysis patients meeting all inclusion/exclusion criteria will be studied in two phases.

In phase 1, subjects will receive a ceiling dose of controlled-release oxycodone hydrochloride (hereafter CR-OC) totaling 40 mg twice daily for 2 weeks prior to the experimental hemodialysis procedure on day 15. Because patients in the hemodialysis group will be anuric, they will undergo hemodialysis three times weekly.10 During that time, they will receive supplemental oral immediate-release oxycodone every 4 h as needed to control their pain up to a visual analog scale level of < 3. These pain levels would correspond with plasma oxycodone concentrations of 20-50 ng/mL.

Patients will be instructed to take their last dose of CR-OC 2 to 3 hours before starting the experimental hemodialysis procedure. This dosing schedule will ensure that the time to CR-OC's maximum concentration (Tmax) and its maximum concentration (Cmax) will be reached at the time of blood sampling at t = 0, enabling accurate assessment of CR-OC's elimination with negligible influence from absorption or redistribution.

At 8:00 am on the 15th day, and this is phase 2 of the study, each individual will undergo hemodialysis for 4 hours. Two independent simultaneous blood samples for measurement of plasma oxycodone concentrations from both arterial inflow (Cin) and venous outflow (Cout) sites will be obtained immediately upon starting hemodialysis (t = 0) and immediately after hemodialysis before shutting off the machine (t = 4). For all calculations and ODE/PDE modeling (see Model Diagram), the oxycodone concentrations from those samples will be combined and averaged. Oxycodone's intradialytic extraction ratio will be calculated from the simultaneously sampled arterial (inflow) and venous (outflow) plasma oxycodone concentrations by dividing their difference by the arterial plasma oxycodone concentrations.

Controls will eat three light meals and a bedtime snack daily. Hemodialysis patients will eat a standard renal diet. Foods will be free of known inhibitors of CYP2D6. Individuals will be digitally abstained from nicotine, caffeine, grapefruit juice and alcohol during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, opioid intolerant Caucasian men and women controls.
* Hemodialysis patients age 44 ± 10 (mean ± SD) years and normal controls 36 ± 9 years.
* No statistically significant difference in weight between hemodialysis and control patients.
* Mean serum creatinine concentrations of 7.29 ± 1.48 mg/dL in hemodialysis patients and 0.81 ± 0.12 mg/dL in controls (normal 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women)
* Mean urine output of 1.83 ± 0.47 mL/hr (44 ± 11 mL/24 hr) in hemodialysis patients and 62.32 ± 16.01 mL/hr (1496 ± 384 mL/24 hr) in controls.
* Patients in both groups with normal liver function. Serum prothrombin time (PT/INR), aPTT, albumin, bilirubin (direct and indirect), liver transaminases, gamma-glutamyl transferase and alkaline phosphatase normal.

Exclusion Criteria:

* In both groups, a clinically significant electrocardiogram (ECG) abnormality.
* An uncontrolled clinically significant cardiovascular condition other than end-stage kidney disease.
* Elevated transaminases, alkaline phosphatase, bilirubin, low phosphodiesterase, elevated ammonia levels, low glucose, elevated lactate, elevated creatinine, and hypoxia (hepatorenal syndrome)
* Serum positive for HIV, hepatitis BsAg, or Hepatitis C
* A history of drug or alcohol abuse within the past 24 months
* Currently participating (or participated within the previous 30 days in an investigational therapeutic or device study
* Female who is pregnant, nursing, or of child-bearing potential not practicing effective contraceptive methods.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Oxycodone's intradialytic mass transfer coefficient | t=0 to t=4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Oscar A Linares, MD, Principal Investigator — Emerio & Lourdes Linares Research and Education Center
Locations (1):
- Oscar A. Linares, MD, Dearborn, Michigan, United States